CLINICAL TRIAL: NCT06402864
Title: Multicenter Randomized Phase III Trial Evaluating Contact X-ray Brachytherapy for Rectal Preservation in Intermediate Substage Rectal Adenocarcinoma
Brief Title: Evaluation Contact X-ray Brachytherapy for Rectal Preservation in Intermediate Substage Rectal Adenocarcinoma
Acronym: TRESOR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-506885-30-00; 2023/3684 (Other: CSET number)
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Adult With Intermediate Low or Mid Rectal Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: It is an open label phase III randomized controlled clinical trial comparing 2 arms:
  * Control arm A consists in TNT regimen, with an induction chemotherapy Modified FOLFIRINOX (mFOLFIRINOX) 6 cycles over 12 weeks, followed by nCRT 50 Gy over 5 weeks with concomitant capecitabine (CAP50 Gy).
  * Experimental arm B consists in addition of three fractions of CXB every two weeks between end of mFOLFIRINOX and nCRT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control arm A (No Intervention): Control arm A consists in TNT regimen, with an induction chemotherapy Modified FOLFIRINOX (mFOLFIRINOX) 6 cycles over 12 weeks, followed by neoadjuvant chemo radiotherapy (nCRT) 50 Gy over 5 weeks with concomitant capecitabine (CAP50 Gy).
- Experimental arm B (Experimental): Experimental arm B consists in addition of three fractions of CXB every two weeks between end of mFOLFIRINOX and nCRT
  Interventions: Radiation: contact X-ray brachytherapy (CXB)

INTERVENTIONS:
Radiation: contact X-ray brachytherapy (CXB) — 3 fractions of contact X-ray brachytherapy (CXB) every two weeks before neoadjuvant chemo radiotherapy (nCRT).
  Arms: Experimental arm B

SUMMARY:
Indication : Adult patients with intermediate low or mid rectal adenocarcinoma to be treated with total neoadjuvant therapy (TNT) potentially eligible for rectal preservation.

Primary objective is to assess efficacy of contact X-ray brachytherapy (CXB) in addition to TNT in order to increase survival with organ preservation (OP), in selected intermediate risk group of rectal adenocarcinomas (size from 3.1 to 6 cm, cT2N1 or T3N0-1, M0).

DETAILED DESCRIPTION:
It is an open label phase III randomized controlled clinical trial comparing 2 arms:

* Control arm A consists in TNT regimen, with an induction chemotherapy Modified FOLFIRINOX (mFOLFIRINOX) 6 cycles over 12 weeks, followed by nCRT 50 Gy over 5 weeks with concomitant capecitabine (CAP50 Gy).
* Experimental arm B consists in addition of three fractions of CXB every two weeks between end of mFOLFIRINOX and nCRT.

Clinical, endoscopic and radiological evaluation will be performed 7 weeks after the end of nCRT in both arms:

* In case of cCR, local excision or surveillance will be proposed to patients regarding center choice
* In the absence of cCR patients will be treated by TME, followed by adjuvant chemotherapy (mFOLFOX 6 cycles or capecitabine 3 cycles over 12 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically proven rectal adenocarcinoma
* Intermediate risk factors: size ≥ 3.1 cm and ≤ 6 cm, < 66% circumference, cT2N1 or T3N0-1, M0 at diagnostic.
* Accessible by digital rectal exam, distal or middle rectum (<11 cm from anal verge), not significantly involving the anal canal (external sphincter not involved) at diagnostic.
* Operable patient
* Patient who is about to start mFolfirinox chemotherapy. The registration is possible before, during or at the end of 4 cycles of mFolfirinox chemotherapy
* Age ≥ 18 years
* WHO status 0 or 1 at diagnosis
* Biological values within the following limits: Total Bilirubin ≤ 1.5 times the upper limit of normal (ULN); ASAT and ALAT ≤ 5 N; Creatinine ≤ 1.5 N and creatinine clearance> 60 ml/min; Neutrophils ≥ 1.5. 109 / L; Platelets ≥ 150. 109 / L; Hemoglobin ≥ 9 g / dL (patients can be included even if they have been transfused); Albuminemia≥30g / L before starting mFolfirinox chemotherapy;
* Women of childbearing potential must have a negative serum β-HCG pregnancy test within 15 days prior to the administration of the first study treatment or urine pregnancy 72 hours prior to the administration of the first study treatment.
* Sexually active women of childbearing potential must agree to use a highly effective method of contraception,
* Sexually actives males patients must agree to use condom during the study and for at least 6 months after the last study treatment administration. Also, it is recommended their women of childbearing potential partner use a highly effective method of contraception for the same duration.
* Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
* Patients must be affiliated to a social security system or beneficiary of the same

Exclusion Criteria:

* Other cancer in the 5 years prior to start m Folfirinox chemotherapy or concomitant (except in situ cancer of the cervix, or basal cell carcinoma of the skin).
* History of pelvic irradiation or pelvis surgery
* Early tumor (T1-2N0, size < 3.1 cm) or advanced tumor (T3 > 6cm of circumference, T4, N2, M1) at diagnostic
* Patient who stopped mFolfirinox after 3 cycles or less
* Dihydropyrimidine dehydrogenase (DPD) deficiency. The blood uracil level must be measured at screening. The uracilemia dosing result is mandatory prior the inclusion of patient.
* Given the oxaliplatin-related risk of prolongation of QT, patient with hypokalemia less than normal, hypomagnesemia, hypocalcemia, and QT/QTc interval longer than 450 msec for men and longer than 470 msec for women on the inclusion ECG should not be allowed at diagnostic.
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV, unstable angina pectoris, history of myocardial infarction in the last 3 months, significant arrhythmia).
* Unbalanced serious illness, underlying infection likely to prevent the patient from receiving treatment current pregnancy (obligatory pregnancy test at baseline) or breastfeeding.
* Psychiatric illness compromising the understanding of information or the conduct of the study.
* Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent.
* Inability to sign informed consent or to undergo medical follow-up of the test for geographical, social or psychological reasons.
* Pregnant or breastfeeding women
* No other anti-tumour prior treatments (chemotherapy, hormone therapy, biologic response inhibitors, targeted therapy) may be used for rectal adenocarcinoma. All live vaccines are prohibited before starting mFolfirinox chemotherapy.
* The combination of warfarin (Coumadine®) with an mFOLFIRINOX regimen, FOLFOX or capecitabine is not recommended. It is preferable to use heparin or LMWH. If warfarin cannot be avoided, more frequent monitoring of prothrombin ratio and INR is necessary.
* Pimozide (Orap®), and cisapride (Prepulsid®) are formally contraindicated: increased risk of ventricular arrhythmias, especially torsades de pointes before starting mFolfirinox chemotherapy
* Known history of hypersensitivity to, fluorouracil, capecitabine, oxaliplatin, irinotecan, folinic acid, or to any of their excipients, according to the SmPCs of these products.
* Recent or concomitant treatment with brivudine, according to the SmPC of fluorouracile and of capecitabine before starting mFolfirinox chemotherapy;
* Chronic inflammatory bowel disease and/or bowel obstruction and in case of concomitant use with St John's Wort, according to the SmPC of irinotecan before starting mFolfirinox chemotherapy;
* Peripheral sensory neuropathy with functional impairment prior to first treatment, according to the SmPC of oxaliplatin before starting mFolfirinox chemotherapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2029-06-15 (Estimated); Study Completion 2030-06-15 (Estimated)

PRIMARY OUTCOMES:
Survival with organ preservation | at the end of the study,15 months after the first inclusion
  defined as a rectum intact, owing to:
  * no radical TME,
  * no locoregional regrowth unless amenable to limited curative (R0) salvage surgery by local excision (LE), and no permanent stoma (including a never reversed protective stoma, or a stoma owing to toxicities and/or poor functional outcomes).

CONTACTS AND LOCATIONS:
Overall Officials: Jérome Durand Labrunie, Dr, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (11):
- France (11):
  - Institut Sainte Catherine, Avignon, France
  - Centre Léon Bérard, Lyon, France
  - Centre de radiotéhrapie Charcot, Lyon, France
  - Hôpital Européen, Marseille, France
  - Centre d'oncologie et de radiothérapie, Mâcon, France
  - Centre de Haute Energie, Nice, France
  - Centre Antoine Lacassagne, Nice, France
  - CHU de Saint Etienne, Saint-Etienne, France
  - Institut de cancérologie de l'Ouest, Saint-Herblain, France
  - Institut Gustave Roussy, Villejuif, France
  - Orlam-Bayard, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No